CLINICAL TRIAL: NCT03860766
Title: Photobiomodulation With Infrared Light-emitting Diode (LED) in Different Doses on Strength Capacities and Functional Performance of Handball Players and Healthy Individuals
Brief Title: Photobiomodulation in Different Doses on Strength Capacities and Functional Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 4.188.366
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Low Level Laser Therapy; Performance; Sport
Keywords: Isokinetic; Electromyography; Physiotherapy; Athletic Performance
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sham Group (G-S) (Sham Comparator): The LED will be positioned across the quadriceps and hamstring bilaterally, however, there will be no light emission. However, the volunteer will perform the strength training protocol.
  Interventions: Other: Photobiomodulation
- 50J Infrared LED Group (G-50J) (Experimental): The LED with a wavelength of 940nm, 50J power, will be applied throughout the quadriceps and hamstrings bilaterally, just before the strength training protocol.
  Interventions: Other: Photobiomodulation
- 240J Infrared LED Group (G-240J) (Experimental): The LED with a wavelength of 940nm, 240J power, will be applied across the quadriceps and hamstrings bilaterally, just before the strength training protocol.
  Interventions: Other: Photobiomodulation
- Progressive dose infrared LED group (G-50-240J) (Experimental): The LED with a wavelength of 940nm, initial energy of 50J with an increment of 38J each week to the final energy of 240J, will be applied throughout extension of the quadriceps and hamstrings bilaterally, immediately prior to the performance of the strength training protocol
  Interventions: Other: Photobiomodulation

INTERVENTIONS:
Other: Photobiomodulation — An LED blanket with 267 infrared lamps with predetermined doses will be used, given a wavelength of 940nm, for 5 weeks, it will be applied by all extension of the quadriceps and hamstrings bilaterally, just before the force training protocol for the groups intervention or simulation for the sham group. Photochemical or photophysical effects are expected from its application.

SUMMARY:
Background: Photobiomodulation has been explored for years, with wide clinical use for wound healing and analgesia in varied orthopedic conditions, but the number of research and clinical use has increased during the last decade. Furthermore, considering the performance, the current literature is conflicting and restricted, with divergences in wavelength, power and energy density applied. Therefore, analyze different doses for a answer in short and long time, associated with capacities of strength, fatigue resistance and functional performance of handball players and healthy individuals becomes necessary. Objective: To analyze the effects of the application of LED photobiomodulation on the capacities of strength, functional efficiency, temperature and fatigue resistance of handball players and healthy individuals. Method: The study sample will be composed of 56 male individuals randomly allocated into four groups: LED 50J (G-50J), LED 240J (G-240J), LED 50-240J (G-50-240J) - progressive dose and Sham (G-S). The volunteers will be submitted to an evaluation of muscle performance and functional performance, metabolic, and physiological evaluation. After initial tests, in five consecutive weeks, the LEDT (940nm - infrared) will be applied to the quadriceps femoris muscle and hamstrings, bilaterally, associated with a muscle strength protocol. After 24 hours of the last application TLED, the tests will be repeated. Seven days after the last intervention will be performed a follow-up. For analysis, normality tests will be used to verify the distribution and adequate statistical tests for the appropriate intra and intergroup comparisons, being considered two factors in the comparisons, time, and group. A significance level of 5% will be adopted.

DETAILED DESCRIPTION:
It is a blinded randomized clinical trial. The volunteers will undergo pre-evaluation, 5 weeks of training associated with the LED application, being distributed in two applications per week, and a re-evaluation 24 hours after the last application, totaling a total of approximately 7 weeks. Thus, on the first day (Pre-test) volunteers will be submitted to anthropometric evaluation and evaluation by bioimpedance for analysis of detailed body composition. Then, the maximum voluntary contraction test (CVM) will be performed on the isokinetic dynamometer, together with the electromyographic evaluation. Before and after the evaluation with the isokinetic dynamometer, thermography will be collected. Still, will be evaluated the vertical jump test after 15 minutes of passive rest.

After the initial evaluations, the researcher will go apply the respective interventions, which consist of applying LEDs all over the quadriceps and hamstring bilaterally, while the sham group (GS) will receive the LED application off, without the emission of light. The application will occur for five weeks and will occur twice weekly, on days spaced for at least 48 hours. The same will be done in conjunction with the lower limb strength training protocol.

The tests performed at the time of pre-application of the LED (Pre-test) will be reapplied in the same order 24 hours after the last application of the interventions. After seven days of the last application, the isokinetic evaluation, electromyography, and vertical jump evaluation will be performed. In addition, at the end of the second and fourth weeks, the volunteer will carry out an evaluation with the isokinetic dynamometer, electromyography, plethysmography, and thermography.

ELIGIBILITY:
Inclusion Criteria:

* Handball players with the participation of at least one official match in the last year and attend 70% of the team's activities during the current season; or
* Healthy individuals;

Exclusion Criteria:

* musculoskeletal injury in the last three months;
* cardiovascular diseases;
* use of anabolic, anti-inflammatory and analgesic drugs 72 hours before the evaluations;
* use of alcohol and illicit drugs during the collection period;

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
difference of maximal voluntary contraction | 3 years
  The study was designed to detect a difference of maximal voluntary contraction between the groups, following the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Girasol, Student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The datas will be sharing in form of manuscript.

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Ferraresi C, Beltrame T, Fabrizzi F, do Nascimento ES, Karsten M, Francisco Cde O, Borghi-Silva A, Catai AM, Cardoso DR, Ferreira AG, Hamblin MR, Bagnato VS, Parizotto NA. Muscular pre-conditioning using light-emitting diode therapy (LEDT) for high-intensity exercise: a randomized double-blind placebo-controlled trial with a single elite runner. Physiother Theory Pract. 2015 Jul;31(5):354-61. doi: 10.3109/09593985.2014.1003118. Epub 2015 Jan 14. PMID 25585514
- [Background] Anders JJ, Lanzafame RJ, Arany PR. Low-level light/laser therapy versus photobiomodulation therapy. Photomed Laser Surg. 2015 Apr;33(4):183-4. doi: 10.1089/pho.2015.9848. No abstract available. PMID 25844681